CLINICAL TRIAL: NCT01906697
Title: The Effect of RF Turbinoplasty Versus Two Other Methods in Management of Polypoid Change of Middle Turbinates: A Randomized Trial.
Brief Title: The Effect of RF Turbinoplasty in Polypoid Change of Middle Turbinates
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Babak Saedi, Associate professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 92--02-48-6933
Record Dates: First submitted 2013-07-19; First posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Nasal Polyposis; Sinusitis
MeSH Terms: conditions — Nasal Polyps; Sinusitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- group B (Active Comparator): middle turbinate resection
  Interventions: Procedure: middle turbinate resection
- group C (Active Comparator): middle turbinate medialization
  Interventions: Procedure: middle turbinate medialization
- group A (Active Comparator): middle turbinate Radio Frequency (RF) turbinoplasty
  Interventions: Procedure: middle turbinate Radio Frequency (RF) turbinoplasty

INTERVENTIONS:
Procedure: middle turbinate Radio Frequency (RF) turbinoplasty — middle turbinate Radio Frequency (RF) turbinoplasty
  Arms: group A
Procedure: middle turbinate resection — middle turbinate resection
  Arms: group B
Procedure: middle turbinate medialization — middle turbinate medialization
  Arms: group C

SUMMARY:
The aim of this study is to evaluate the effect of middle turbinate Radio Frequency (RF) turbinoplasty with middle turbinate resection and medialization

DETAILED DESCRIPTION:
The management of middle turbinate in treatment of nasal polyposis is still an interesting debatable topic. The surgical access and its possible role in pathophysiology of sinusitis are two important points about its treatment. On the one hand, middle turbinate resection can improve surgical access and possibly reduce the nasal polyposis recurrence. On the other hand, there are some reports of anosmia, empty nose syndrome, synechia, and difficulties in revision surgery. Also, synechia, lateralization, and possibly recurrence can be the possible outcome after middle turbinate preservation.

Among different modalities, radiofrequency (RF) gradually increase its popularity as surgical tools, which can treat mucosal hypertrophy without any tissue removal. Inferior turbinate is a famous place for its usage, especially for decreasing of the nasal obstruction. Also, some authors have showed its effect on refractory allergic rhinitis, which is not only related to reducing of nasal obstruction, but also it is related to changing of the allergic mediators. [5, 6] Comparing to other treatments for turbinates is sparing its overlaid mucosa, which can reduce the possible future morbidities.

Probably considering of the above mention points, RF has a possible impact on the polypoid changes of middle turbinates and possibly does not have the same deleterious effect of the resection on cilia of mucosal layer. Therefore, we performed a randomized clinical trial to compare its outcome with two famous methods of the middle turbinate management: partial resection and medialization.

ELIGIBILITY:
Inclusion Criteria:

The patients with sinusitis who suffered from nasal polyposis which was resistant to maximal medical treatment (i.e. one puff of Fluticasone nasal spray twice daily plus amoxicillin clavulanic acid 625 mg tablet three times daily, for at least one month ).

Exclusion Criteria:

* floppy' change of the middle turbinate in the end of surgery.
* systemic disease (e.g. hypertension, Wegener's granulomatosis, cystic fibrosis or sarcoidosis),
* immune suppression,
* revision surgery,
* counter-indications for any of the postoperative drug usage (e.g. diabetes or pregnancy), or
* any type of septoplasty indications are excluded from this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-09 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
The Sino-Nasal Outcomes Test 22 | three months after surgery
  The Sino-Nasal Outcome Test-22 (SNOT-22) questionnaire is a disease-specific questionnaire involving 22 symptoms combining rhinologic issues with general health issues.
The Sino-Nasal Outcomes Test 22 | 6 months after surgery
  The Sino-Nasal Outcome Test-22 (SNOT-22) questionnaire is a disease-specific questionnaire involving 22 symptoms combining rhinologic issues with general health issues.
The Sino-Nasal Outcomes Test 22 | one year after surgery
  The Sino-Nasal Outcome Test-22 (SNOT-22) questionnaire is a disease-specific questionnaire involving 22 symptoms combining rhinologic issues with general health issues.

CONTACTS AND LOCATIONS:
Overall Officials: Babak Saedi, professor, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, Tehran, Tehran Province, Iran